CLINICAL TRIAL: NCT06345716
Title: Paracetamol-Tramadol and Paracetamol-caffeine Versus Placebo in the Emergency Discharge Treatment of Renal Colic
Acronym: RC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, PROFESSOR, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: renal colic 2024
Record Dates: First submitted 2024-03-08; First posted 2024-04-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Renal Colic
Keywords: renal colic; paracetamol-tramadol; paracetamol-cafeine; placebo
MeSH Terms: conditions — Renal Colic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Paracétamol-tramadol (Experimental): Each patient received 1 tablet * 2/day synalvic (325 mg of paracetamol + 37.5 mg of tramadol) for 7 days.
  Interventions: Drug: paracétamol tramadol
- Paracetamol-caffeine (Experimental): Each patient received 1 tab * 3/d stopalgic extra (65mgcaffeine+500mg paracetamol) for 7 days
  Interventions: Drug: Paracétamol cafeine
- Placebo (Experimental): Each patient received 1 tab * 3 / d of placebo (flour) every day for 7 days.
  *For the three groups, the tablets were packaged hermetically in identical envelopes taken at random to respect double blinding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: paracétamol tramadol — Each patient received 1 tablet * 2/day synalvic (325 mg of paracetamol + 37.5 mg of tramadol) for 7 days
  Other Names: B
  Arms: Paracétamol-tramadol
Drug: Paracétamol cafeine — Each patient received 1 tab * 3/d stopalgic extra (65mgcaffeine+500mg paracetamol) for 7 days
  Other Names: A
  Arms: Paracetamol-caffeine
Drug: Placebo — Each patient received 1 tab * 3 / d of placebo (flour) every day for 7 days
  Other Names: C
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, single-blind study. Patients included in the study after successful treatment of the acute attack were randomized upon discharge from the Emergency Department into three groups: oral paracetamol-tramadol group, oral paracetamol-caffeine group and oral placebo group.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blind study. Patients included in the study after successful treatment of the acute attack were randomized upon discharge from the Emergency Department into three groups: oral paracetamol-tramadol group, oral paracetamol-caffeine group and oral placebo group.

Different parameters are collected on a standard form prepared for all cases of renal colic included in our study. This sheet essentially contains:

Temperature, systolic and diastolic blood pressure, heart rate, pain intensity assessed by VAS, abdominal tenderness as well as the existence of Giardano signs.

Additional examinations were not systematically carried out for all patients: AUSP, ECBU, renal ultrasound, creatinemia and blood sugar. Their realization depended on the clinical context.

The use of imaging was done following the indications specified in the text of the consensus of the French Society of Emergency Medicine (updated in 2008)

ELIGIBILITY:
Inclusion Criteria:

* -Age > 18 years old.
* Consent to participate in the study.
* Pain in the flank/lumbar fossa of sudden onset with urine strips and/or imaging corresponding to the diagnosis of renal colic.
* Pain score at discharge < 30 (visual analog scale - VAS or verbal numerical scale - VAS from 0 to 100).

Exclusion Criteria:

* -Inability to appreciate pain according to the VAS.
* Pregnant or breastfeeding woman.
* Renal insufficiency with creatinine clearance < 60 ml/min.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of RC and ED readmission | 7 day after inclusion
  included recurrence of RC and ED readmission within 7-day follow-up

SECONDARY OUTCOMES:
mean time interval | 7 day after inclusion
  mean time to recurrence of pain
side effects | 7 days 30 days
  occurence of side effects

OTHER OUTCOMES:
Adverse effects | 7 days 30 days
  -Adverse effects of treatment and its tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Khaoula Bel Haj Ali, Study Director — CHU Fattouma Bourguiba Monastir, service des urgences
Locations (1):
- Semir Nouira, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No